CLINICAL TRIAL: NCT04732975
Title: Mason Heart Study With Magnetocardiography
Brief Title: Mason Heart Study With MCG
Acronym: MHS-MCG
Status: Suspended | Type: Observational
Why Stopped: Resourcing
Sponsor: Genetesis Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1000-3
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Acute Myocardial Injuries
Keywords: ischemia; acute myocardial injuries; CardioFlux; Cardiovascular disease; MCG
MeSH Terms: conditions — Ischemia; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: CardioFlux — Non-invasive screening for ACS

SUMMARY:
Heart disease is the number one cause of death in the United States, with over 650,000 deaths in 2019 alone. Many healthy individuals possess key risk factors for heart disease which include but are not limited to high blood pressure, high cholesterol, family history of heart disease, and diabetes. The Mason Heart Study-MCG (MHS-MCG) registry is designed to collect magnetocardiography (MCG) scans on a select group of healthy volunteers who work for the city of Mason, OH, with and without cardiac symptoms, illnesses, and/or risk factors. CardioFlux is used as a noninvasive MCG tool that analyzes and records the magnetic fields of the heart to detect various forms of heart disease. There will be a 12-month duration of the study where we propose to collect screening data from approximately 250 volunteers who present to the Genetesis facility for a 5-minute CardioFlux MCG scan. The volunteers will be contacted at intervals over a 1-year period for follow-up data and may choose whether or not they would like to provide follow-up data or participate in another scan.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of enrollment.

Exclusion Criteria:

1. < 18 years of age
2. Patients unable to fit into device
3. Non-ambulatory patients
4. Positive response on CardioFlux Pre-Screening Form
5. Patients with claustrophobia or unable to lie supine for 5 minutes
6. Pregnant women
7. Poor candidate for follow-up (e.g. no access to phone)
8. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All healthy and non-healthy individuals who are 18 or older.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
specificity and accuracy statistics | 6 months
  analyzing the specificity and accuracy of CardioFlux

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Senagore, M.D., Principal Investigator — Genetesis Inc.
Locations (1):
- Genetesis Facility, Mason, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaikovsky I, Hailer B, Sosnytskyy V, Lutay M, Mjasnikov G, Kazmirchuk A, Bydnyk M, Lomakovskyy A, Sosnytskaja T. Predictive value of the complex magnetocardiographic index in patients with intermediate pretest probability of chronic coronary artery disease: results of a two-center study. Coron Artery Dis. 2014 Sep;25(6):474-84. doi: 10.1097/MCA.0000000000000107. PMID 24667125
- [Background] Goernig M, Liehr M, Tute C, Schlosser M, Haueisen J, Figulla HR, Leder U. Magnetocardiography based spatiotemporal correlation analysis is superior to conventional ECG analysis for identifying myocardial injury. Ann Biomed Eng. 2009 Jan;37(1):107-11. doi: 10.1007/s10439-008-9598-5. Epub 2008 Nov 18. PMID 19015988
- [Background] Hailer B, Chaikovsky I, Auth-Eisernitz S, Schafer H, Van Leeuwen P. The value of magnetocardiography in patients with and without relevant stenoses of the coronary arteries using an unshielded system. Pacing Clin Electrophysiol. 2005 Jan;28(1):8-16. doi: 10.1111/j.1540-8159.2005.09318.x. PMID 15660796
- [Background] Kwong JS, Leithauser B, Park JW, Yu CM. Diagnostic value of magnetocardiography in coronary artery disease and cardiac arrhythmias: a review of clinical data. Int J Cardiol. 2013 Sep 1;167(5):1835-42. doi: 10.1016/j.ijcard.2012.12.056. Epub 2013 Jan 19. PMID 23336954
- [Background] Lim HK, Kwon H, Chung N, Ko YG, Kim JM, Kim IS, Park YK. Usefulness of magnetocardiogram to detect unstable angina pectoris and non-ST elevation myocardial infarction. Am J Cardiol. 2009 Feb 15;103(4):448-54. doi: 10.1016/j.amjcard.2008.10.013. Epub 2008 Dec 25. PMID 19195500